CLINICAL TRIAL: NCT04433156
Title: A Single Arm, Multi-center, Phase II Clinical Trial of VR-CAP in the First-line Treatment for Patients With Marginal Zone Lymphoma
Brief Title: VR-CAP in the First-line Treatment for Patients With Marginal Zone Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yanyan Liu, Director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNSZLYYNHL03
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Marginal Zone Lymphoma
Keywords: Marginal Zone Lymphoma; VR-CAP
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Bortezomib; Rituximab; Epirubicin; Cyclophosphamide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR-CAP (Experimental): Rituximab, 375 mg/m2, Intravenous administration on day 0, Bortezomib, 1.3 mg/m2 hypodermic injection on day 1 and 4, combined with regimen: Cyclophosphamide, Epirubicin, and Prednisone: repeated every 3 weeks, up to 6 cycles.
  Interventions: Drug: Bortezomib; Drug: Rituximab; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Prednisone

INTERVENTIONS:
Drug: Bortezomib — 1.3 mg/m2, hypodermic injection on day 1 and day 4 of each 3-week cycle until disease progression/stable disease after 2/4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Bortezomib Injection
Drug: Rituximab — 375 mg/m2, Intravenous administration on day 0 of each 3-week cycle until disease progression/stable disease after 2/4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: RiTUXimab Injection
Drug: Epirubicin — 70 mg/m2, Intravenous administration on day 1 of each 3-week cycle until disease progression/stable disease after 2/4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Epirubicin hydrochloride
Drug: Cyclophosphamide — 750 mg/m2, Intravenous administration on day 1 of each 3-week cycle until disease progression/stable disease after 2/4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Cyclophosphamide Injection
Drug: Prednisone — 100mg, oral administration on day 1 to 5 of each 3-week cycle until disease progression/stable disease after 2/4 cycles treatment or unacceptable toxicity develops, up to 6 cycles
  Other Names: Prednisone Oral Product

SUMMARY:
This is a prospective single arm, multi-center, phase II clinical trial to observe the efficacy and safety of VR-CAP (Bortezomib and Rituximab-Cyclophosphamide, Epirubicin and Prednisone) in the first-line treatment for patients with marginal zone lymphoma.

DETAILED DESCRIPTION:
Marginal zone lymphoma (MZL) is a relatively common group of non-Hodgkin's lymphoma (NHL). The incidence rate is only inferior to diffuse large B cell lymphoma (DLBCL) and follicular lymphoma (FL). Currently, NCCN guidelines recommend same treatment plan of FL like R-CHOP as the primary treatment for MZL. However, due to the great difference in cell origin and biological characteristics between FL and MZL, some patients can not achieve complete remission or relapse quickly after standard first-line treatment. A number of phase II clinical studies have evaluated the good efficacy of rituximab combined with chemotherapy in the treatment of MZL. Previous studies have shown that NF-κB signaling pathway is in abnormal activation state in MZL. Bortezomib, a proteasome inhibitor targeting NF-κB pathway, has a promising therapeutic prospect in relapsed and refractory MZL. The goal of our trial is to assess the efficacy and safety of VR-CAP (Bortezomib and Rituximab-Cyclophosphamide, Epirubicin and Prednisone) in the first-line treatment for patients with marginal zone lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 70 years old (including 18 and 70)
2. Diagnosed as marginal zone lymphoma
3. No receiving chemotherapy before enrollment
4. Indications for treatment: 1) symptoms related to tumor; 2) end-organ function damage; 3) large mass; 4) continuous or rapid progress of disease; 5) patient's willingness
5. Having at least one measurable lesions
6. World health organization-Eastern Cooperative Oncology Group Performance tatus (ECOG) 0-1
7. Life expectancy no less than 3 months
8. enough main organ function
9. Pregnancy test within 7 days must be negative for women of childbearing period, and appropriate measures should be taken for contraception for women in childbearing period during the study and six months after this study
10. Agreeing to sign the written informed consents

Exclusion Criteria:

1. Diagnosed as central nervous system lymphoma
2. World health organization-Eastern Cooperative Oncology Group Performance tatus (ECOG) ≥2
3. Other malignant tumor history or active malignant tumor need be treated
4. Serious surgery and trauma less than two weeks
5. Systemic therapy for serious acute/chronic infection
6. Congestive heart failure, uncontrolled coronary heart disease, arrhythmia and heart infarction less than 6 months
7. Active tuberculosis. Patients suspected of active TB need to be examined for chest X-ray, sputum and clinical symptoms and signs
8. HIV-positive, AIDS patients and untreated active hepatitis（HBV/HBV and HCV）
9. Patients with a history of deep vein thrombosis or pulmonary embolism less than 12 months
10. Patients with a history of mental illness
11. Researchers determine unsuited to participate in this trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-04-22 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | from the beginning day of the first cycle (each cycle is 21 days) of treatment to the date of confirmed progressive disease or death, whichever occurs first, up to 2 years after last patient's enrollment
  the total proportion of patients with no progression from date of the first day of treatment to the date of confirmed progressive disease or death which one occurs first

SECONDARY OUTCOMES:
objective response rate | every 6 weeks from the beginning day of the first cycle (each cycle is 21 days) of induction chemotherapy treatment and every 8 weeks from the day of the first cycle of maintenance treatment to 18 months after last patient's enrollment
  the total proportion of patients with complete response (CR) and partial response (PR)
overall survival | from the beginning day of the first cycle (each cycle is 21 days) of treatment to the date of death from any cause, assessed up to 5 years
  from date of first day of treatment to the date of death by any cause
incidence and relationship with study drugs of grade 3-4 adverse events | from the beginning day of the first cycle (each cycle is 21 days) of treatment to 6 months after last patient's enrollment
  the incidence and relationship with study drugs of grade 3 or 4 adverse events (based on NCI CTC-AE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Liu, M.D. Ph.D, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No